CLINICAL TRIAL: NCT02494050
Title: Telemedicine for Women With Anhedonia in Bipolar and Unipolar Disorder: Patient Preferences and Outcomes
Brief Title: Telemedicine for Women With Anhedonia in Bipolar and Unipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jacqueline Gollan, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00200085
Record Dates: First submitted 2015-06-30; First posted 2015-07-10 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Depression; Bipolar Disorder; Anhedonia
Keywords: Depression; Bipolar Disorder; Anhedonia; Women
MeSH Terms: conditions — Depression; Bipolar Disorder; Anhedonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Behavioral Activation-Full (Experimental): Twelve weekly sessions of phone therapy using Behavioral Activation Treatment for Anhedonia.
  Interventions: Behavioral: Behavioral Activation-Full
- Behavioral Activation-Short (Experimental): Eight weekly sessions of phone therapy using Behavioral Activation Treatment for Anhedonia.
  Interventions: Behavioral: Behavioral Activation-Short
- Bipolar Disorder Collaborative Care (Active Comparator): Twelve weekly sessions of phone therapy using BDCC manual adapted for anhedonia.
  Interventions: Behavioral: Bipolar Disorder Collaborative Care

INTERVENTIONS:
Behavioral: Behavioral Activation-Full — Behavioral Activation proposes that symptom reduction occurs via monitoring daily activities to identify patterns of low reward and mood, assessing and assigning tasks that generate pleasure and competence, understanding and reducing unproductive avoidance, and improving skill deficits to promote action towards treatment goals.
  Arms: Behavioral Activation-Full
Behavioral: Behavioral Activation-Short — Behavioral Activation proposes that symptom reduction occurs via monitoring daily activities to identify patterns of low reward and mood, assessing and assigning tasks that generate pleasure and competence, understanding and reducing unproductive avoidance, and improving skill deficits to promote action towards treatment goals.
  Arms: Behavioral Activation-Short
Behavioral: Bipolar Disorder Collaborative Care — This manualized treatment focuses on social support and educating patients about medication compliance. The primary focus is to strengthen the patients' self-management skills with education; supporting the clinician's decision making using practice guidelines; enhancing access to care, continuity of care, and information flow through the use of the clinician.
  Arms: Bipolar Disorder Collaborative Care

SUMMARY:
Anhedonia, characterized as (a) the diminished motivation to participate in activities, and/or (b) diminished enjoyment of a pleasurable activity are common symptoms among women diagnosed with mood disorders. This trial aims to test three treatments adapted to reduce anhedonia.

The investigators will compare three treatment groups, specifically, two doses of Behavioral Activation treatment for anhedonia (i.e., 12 weeks vs. 8 weeks of BA) with an active comparator treatment, Bipolar Disorder Collaborative Care (12 weeks of BDCC). BA is a psychotherapy approach that helps participants to identify and modify environmental sources of their depression. BDCC is a supportive care approach that educates participants to optimize their medication initiation or their existing medication regimen. The time frame for this study will be between 12-14 weeks. Specifically, participants will be evaluated and enrolled within one week, then received up to 12 weeks of treatment (tracked through this time) and then complete two evaluations (one at week 8) and another at the end of treatment (an expected average of 12-14 weeks after enrolling into treatment).

Primary analyses aim to compare the dose-mechanism change in BA relative to a standard medication optimizing protocol, BDCC. The secondary analyses are to evaluate individual differences in stated patient preferences for treatment, and group differences in treatment effect on anhedonia, side effects, and quality of life.

DETAILED DESCRIPTION:
Prospective volunteers will be screened by phone and, if eligible, invited to a clinical evaluation in the laboratory, located at Northwestern University. At the laboratory, prospective volunteers complete written informed consent and learn about the study.

All evaluations will measure the following variables: Anhedonia will be assessed using the Snaith-Hamilton Pleasure Scale, Temporal Experience of Pleasure Scale, and Effort-Expenditure for Rewards Task; Mood symptoms will be assessed by the Structured Clinical Interview for DSM-IV, Inventory of Depressive Symptomatology-Clinician Version, Clinician-Administered Rating Scale for Mania, Inventory of Depressive Symptomatology-Clinician version, and Columbia Suicide Severity Rating Scale. Treatment preferences will measured with the Stated Preferences Inventory for Bipolar Disorder. The presence of side effects from medications will be evaluated using the Frequency, Intensity, and Burden of Side Effects measure. Maternal function will be evaluated using the Barkin Index of Maternal Function self-report. Behavioral Inhibition System/Behavioral Activation System and the Behavioral Activation for Depression Scale are used to evaluate activation levels. Reward processing will be measured using the Monetary Incentive Delay Task on the computer and the Reward Probability Index questionnaire.

Enrollment is determined on a set of criteria, whereby participants will be randomized into one of three treatment groups using a computerized randomized number generator using a 1:1:1 ratio. Allocation concealment will be set up so the person enrolling the participant will not know in advance which treatment the participant will receive. Moreover, evaluators will remain blind to treatment assignment. Participants are randomized to receive one of three treatments: 12 weeks of BA, 8 weeks of BA with option to add 4 weeks, and 12 weeks of BDCC. Participants are asked to participate in two follow-up evaluations at the laboratory, scheduled at Weeks 8 and 12. The study ends after the Week 12 evaluation (approximately 12-14 weeks after enrolling into the treatment).

ELIGIBILITY:
Inclusion Criteria:

* Currently experiencing a score ≥ 20 on a clinician-administered scale of anhedonia
* Currently experiencing two or more symptoms of depression with bipolar disorder either Type I or II (one of these symptoms should be anhedonia) OR
* Currently experiencing two or more symptoms of unipolar depression, without current psychotic features (one of these symptoms should be anhedonia)
* Currently on a medication for a mood disorder
* Proficiency in English
* Able to provide informed consent

Exclusion Criteria:

* Current psychosis (schizoaffective, schizophreniform, delusional disorder)
* Current suicide risk sufficient to preclude treatment on an outpatient basis
* Severe, unstable concurrent psychiatric conditions likely to require hospitalization within six months (ex. hazardous substance use evidenced by a score > 10 on the Alcohol Use Disorders Identification Test or > 2 on the Drug Use Disorders identification Test)
* Current incarcerated or on probation due to criminal allegations
* Currently pregnant
* Cognitive impairment
* Those living in the United States on a VISA
* Those currently in psychotherapy

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Snaith-Hamilton Pleasure Scale-Clinician Version | approximately 12-14 weeks after enrolling into the treatment
  Clinician-administered measure of anhedonia spanning the domains of: interests, social interaction, sensory experience, and food/drink.

SECONDARY OUTCOMES:
Inventory of Depressive Symptomatology-Clinician | approximately 12-14 weeks after enrolling into the treatment
  Clinician-administered measure of depression severity
Clinician-Administered Rating Scale for Mania | approximately 12-14 weeks after enrolling into the treatment
  Clinician-administered measure of the severity of manic symptoms which includes items that focus on Bipolar and items that focus on psychosis

CONTACTS AND LOCATIONS:
Overall Officials: Jackie K Gollan, Ph.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided